CLINICAL TRIAL: NCT00614718
Title: Failure of Chronically Implanted Defibrillator Leads -Incidence and Management A Retrospective Multicenter Study
Brief Title: Failure of Chronically Implanted Defibrillator Leads -Incidence and Management
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Christian Sticherling, MD, University Hospital Basel, Division of Cardiology
Other Study IDs: USB01
Record Dates: First submitted 2008-01-30; First posted 2008-02-13 (Estimated); Last update posted 2008-02-13 (Estimated); Status verified 2008-01

CONDITIONS: Death, Sudden, Cardiac; Ventricular Fibrillation
Keywords: Implantable cardioverter defibrillator; lead failure; pace/sense lead; ICD complication; inappropriate therapy; Defibrillators
MeSH Terms: conditions — Death, Sudden, Cardiac; Ventricular Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Total number of patients receiving an ICD between 1993 and 2004 and not having re interventions due to malfunctioning leads.
- 2: Patients with ICD lead failure receiving a new ICD lead
- 3: Patients with ICD lead failure but intact shock-coil of the ICD lead receiving only an additional pace/sense lead.

SUMMARY:
Comparison of two different approaches to address the problem of malfunctioning ICD-leads. These leads consist of two parts. One that is used for detection of arrhythmias(and pacing if required) (Pace/Sense) and a second part that is used to deliver therapy is needed (Shock-coil).

The two approaches compared are:

Replacement of the entire lead in case of any lead malfunction versus placement of an additional pace/sense-lead if the shock-coil of the exiting lead was still functional.

DETAILED DESCRIPTION:
Therapy with an implantable cardioverter defibrillator (ICD) has become a standard treatment for an increasing number of patients suffering from different types of heart diseases which can lead to fatal arrhythmias. This therapy was established about 20 Years ago and malfunctioning electrodes of these devices have been, and still are a serious problem leading to inappropriate therapy (shocks)or missed live saving therapy.

In case of a malfunctioning electrode it is established clinical practice to either replace the entire ICD electrode (which is used for detecting the arrhythmias as well as delivering the shock) or just to implant an additional electrode for detection of the arrhythmia (and pacing if required) given that the "shock"-part of the existing electrode is still functional.

There is no longterm outcome data comparing these two strategies. We included 1317 consecutive patients with an ICD implanted at three European centers between 1993 and 2004. Incidence of lead failure, type of lead used, approach and outcome were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Implantation of an ICD between 1993 and 2004

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1317 consecutive patients with an ICD implanted at three European centers between 1993 and 2004
Sampling Method: Non-Probability Sample
Enrollment: 1317 (Actual)
Dates: Start 1993-01; Primary Completion 2004-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Time to lead failure or lead failure recurrence | from inclution to death or end of follow up (Jan 2004)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Sticherling, MD, Principal Investigator — University Hospital Basel, Dept. Cardiology
Locations (3):
- Germany (2):
  - Herzzentrum Bad Krozingen, Bad Krozingen
  - Benjamin Franklin, Division of Cardiology,, Berlin
- University Hospital, Basel, Switzerland